CLINICAL TRIAL: NCT04645797
Title: A Phase 1 Dose Escalation Study to Evaluate Safety, Tolerability, and Pharmacokinetics/ Pharmacodynamics of APR003 in Patients With Advanced Colorectal Cancer (CRC) With Malignant Liver Lesions
Brief Title: A Dose Escalation Study of APR003 in Patients With Advanced Colorectal Cancer (CRC) With Malignant Liver Lesions
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated prematurely due to internal corporate decision
Sponsor: Apros Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APR003-001
Record Dates: First submitted 2020-09-16; First posted 2020-11-27 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Advanced Colorectal Carcinoma

STUDY DESIGN:
Intervention Model Description: Phase 1 Dose Escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- APR003 Dose Escalation (Experimental): This portion of the study will evaluate the safety and pharmacokinetics of a range of APR003 doses administered once a week for 21 days in subjects with advance colorectal cancer (CRC) with metastases to the liver and to determine the RP2D.
  Interventions: Drug: APR003

INTERVENTIONS:
Drug: APR003 — This portion of the study further explores the clinical activity, safety, pharmacokinetics and pharmacology of APR003 monotherapy at the RP2D and to assess the antitumor activity of APR003 in subjects with unresectable CRC with liver metastases.

SUMMARY:
A Phase 1 dose escalation study to evaluate APR003 in patients with advanced colorectal cancer (CRC) with malignant liver lesions

DETAILED DESCRIPTION:
APR003 is a small molecule TLR7 agonist that concentrates in the GI, and liver with limited systemic exposure. It is designed to increase the therapeutic window of a TLR7 agonist by minimizing the side-effects associated with generalized systemic immune activation and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0 or 1
* Must have disease that is considered non-surgically resectable.
* Relapsed or persistent/refractory to at least two prior systemic treatment regimens for locally advanced or metastatic disease considered to be standard-of-care (SOC).
* Must have previously received an irinotecan or oxaliplatin-based therapy, as well as a targeted antibody therapy for metastatic disease
* Tumors that are MSI-H/dMMR must have previously received checkpoint inhibitor therapy
* Adequate hepatic function
* Adequate renal function
* Normal coagulation panel
* Willingness to use effective contraception

Exclusion Criteria:

* Current or history of CNS metastases
* Significant cardiovascular disease
* Pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2022-05-07 (Actual); Study Completion 2022-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Weitzman, MD, Study Director — Apros Therapeutics, Inc; Trinh Le, Study Director — Apros Therapeutics, Inc
Locations (4):
- United States (4):
  - AdventHealth Orlando, Orlando, Florida
  - Carolina BioOncology Institute Cancer Research Clinic, Huntersville, North Carolina
  - NEXT Oncology - Austin, Austin, Texas
  - NEXT Oncology - San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller A, Le T, Holland J, et al1167 APR003, an oral liver- and GI-targeted TLR7 agonist, elicits a robust type I interferon response in advanced colorectal cancer patientsJournal for ImmunoTherapy of Cancer 2022;10:doi: 10.1136/jitc-2022-SITC2022.1167

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort -1: 25 MG once a week for 21 days in subjects with advance colorectal cancer (CRC) with metastases to the liver and to determine the RP2D.
- Cohort 1: 50 MG once a week for 21 days in subjects with advance colorectal cancer (CRC) with metastases to the liver and to determine the RP2D.
- Cohort 2: 100 MG once a week for 21 days in subjects with advance colorectal cancer (CRC) with metastases to the liver and to determine the RP2D.
- Cohort 3: 175 MG once a week for 21 days in subjects with advance colorectal cancer (CRC) with metastases to the liver and to determine the RP2D.
- Cohort 4: 250 MG once a week for 21 days in subjects with advance colorectal cancer (CRC) with metastases to the liver and to determine the RP2D.
- Cohort 5: 350 MG once a week for 21 days in subjects with advance colorectal cancer (CRC) with metastases to the liver and to determine the RP2D.
- Cohort 6: 500 MG once a week for 21 days in subjects with advance colorectal cancer (CRC) with metastases to the liver and to determine the RP2D.
Period: Overall Study
Arm/Group | Cohort -1 | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Started | 6 | 4 | 1 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 4 | 1 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 3 | 3 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 3 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort -1: 25 MG once a week
- Cohort 1: 50 MG once a week
- Cohort 2: 100 MG once a week
- Total: Total of all reporting groups
Arm/Group | Cohort -1 | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 6 | 4 | 1 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 1 | 10
  >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Median (Full Range); unit: years] | 50.5 [47 to 74] | 52 [51 to 64] | 52 [52 to 52] | 52 [47 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 3
  Male | 4 | 4 | 0 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 3 | 1 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 4 | 0 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — All patients enrolled in United States
  participants
    United States | 6 | 4 | 1 | 11
ECOG Performance Status [Median (Full Range); unit: units on a scale] — Eastern Cooperative Oncology Group (ECOG) performance status was a 6-level item used to assess the physical health of participants and ranged from 0 (fully active), 1 (restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature) to 5 (dead).
  units on a scale | 1 [0 to 1] | 0.5 [0 to 1] | 0 [0 to 0] | 1 [0 to 1]
Stage at Trial Entry [Count of Participants; unit: Participants] — Tumor stage at trial entry was classified according to the American Joint Committee on Cancer (AJCC) 8th Edition staging system. All participants had Stage IV disease, with substages distributed as follows: IVB, IV, and IVC. Higher stage substages indicate more advanced disease.
  Participants
    IVB | 2 | 4 | 1 | 7
    IV | 2 | 0 | 0 | 2
    IVC | 2 | 0 | 0 | 2
Current Stage-Tumor (T) [Count of Participants; unit: Participants] — Current Tumor (T) stage at trial entry was assessed according to the AJCC 8th Edition staging system. The substages ranged from T2 through T4a, with higher T categories indicating larger tumor size and/or greater local invasion.
  Participants
    T2 | 1 | 0 | 0 | 1
    T3 | 5 | 1 | 0 | 6
    T4a | 0 | 2 | 0 | 2
    T4 | 0 | 0 | 1 | 1
    Unknown | 0 | 1 | 0 | 1
Current Stage-Metastasis (M) [Count of Participants; unit: Participants] — Current Metastasis (M) stage at trial entry was assessed according to the AJCC 8th Edition staging system. Only patients with M1 and M1b disease were enrolled, representing the presence of distant metastases. Higher M categories indicate more extensive metastatic spread.
  Participants
    M1b | 4 | 4 | 1 | 9
    M1 | 2 | 0 | 0 | 2
Primary Tumor Location [Count of Participants; unit: Participants]
  Colon, Left | 0 | 1 | 1 | 2
  Colon, Right | 0 | 1 | 0 | 1
  Rectal | 2 | 1 | 0 | 3
  Other | 4 | 1 | 0 | 5
Colorectal Type [Count of Participants; unit: Participants]
  Adenocarcinoma | 5 | 4 | 1 | 10
  Mucinous | 1 | 0 | 0 | 1
Grade at Study Entry [Count of Participants; unit: Participants] — Tumor grade at study entry was assessed using standard histopathologic criteria. Enrolled patients included those with Grade 1 (G1), Grade 2 (G2), Grade X (GX; undetermined grade), and unknown grade. Lower grades (G1) generally indicate well-differentiated tumors with better prognosis, while higher grades indicate poorer differentiation and more aggressive disease.
  Participants
    G2 | 5 | 1 | 1 | 7
    GX (grade not assessed) | 1 | 1 | 0 | 2
    G1 | 0 | 1 | 0 | 1
    Unknown | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Determine the Number of Patients With Dose Limiting Toxicities (DLTs)
Description: Determine the number of patients who have experienced a Dose Limiting Toxicities (DLT) evaluated by the investigator based on CTCAE Severity Grade.
Time Frame: Until disease progression, or up to approximately 15 months and 18 days, whichever is first
Measure: Number; unit: participants
Arm/Group | Cohort -1 | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 4 | 1
participants | 0 | 0 | 1

2. Primary Outcome: Maximum Concentration (Cmax) of APR003
Description: Plasma concentration of APR003 was analyzed by a validated liquid chromatography-tandem mass spectrometry assay. Standard PK parameters were determined using non-compartmental methods.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 (Cycle duration is 21 days)
Population: One patient in Cohort 1 was dose-reduced after the first dose from 50 MG to 25 MG and was included only in the Cycle 1 Day 1 analysis. The only patient in Cohort 2 was not analyzed due to incomplete blood collection.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort -1 | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 4 | 0
ng/mL
  Cycle 1 Day 1 | 224 (124) | 158 (85.4) |
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 3 | 0
  Cycle 1 Day 15 | 362 (150) | 148 (85.4) |
  Cycle 2 Day 1: number analyzed (Participants) | 6 | 3 | 0
  Cycle 2 Day 1 | 217 (157) | 121 (65.3) |

3. Primary Outcome: Time-to-maximum Concentration (Tmax) of APR003
Description: as for outcome 2
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 (Cycle duration is 21 days)
Population: as for outcome 2
Measure: Mean (Full Range); unit: hr
Arm/Group | Cohort -1 | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 4 | 0
hr
  Cycle 1 Day 1 | 0.750 [0.5 to 2] | 2.00 [0.5 to 2] |
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 3 | 0
  Cycle 1 Day 15 | 1.00 [0.5 to 1] | 2.00 [1 to 4] |
  Cycle 2 Day 1: number analyzed (Participants) | 6 | 3 | 0
  Cycle 2 Day 1 | 1 [0.5 to 4] | 2.00 [2 to 4] |

4. Primary Outcome: Area Under the Curve (AUC) From Time Zero to 24 hr (AUC0-24) of APR003
Description: as for outcome 2
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15 (Cycle duration is 21 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort -1 | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 4 | 0
ng*hr/mL
  Cycle 1 Day 1 | 597 (209) | 489 (137) |
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 2 | 0
  Cycle 1 Day 15 | 862 (355) | 412 (89) |

5. Primary Outcome: AUC From Time Zero to Time Infinity (AUC0-ꝏ) of APR003
Description: as for outcome 2
Time Frame: Cycle 1 Day 1 (Cycle duration is 21 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort -1 | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 4 | 0
ng*hr/mL | 601 (212) | 497 (134) |

6. Primary Outcome: AUC Over the Dosing Interval (AUClast) of APR003
Description: as for outcome 2
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 (Cycle duration is 21 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort -1 | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 4 | 0
ng*hr/mL
  Cycle 1 Day 1 | 597 (209) | 489 (137) |
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 3 | 0
  Cycle 1 Day 15 | 830 (330) | 443 (112) |
  Cycle 2 Day 1: number analyzed (Participants) | 6 | 3 | 0
  Cycle 2 Day 1 | 525 (370) | 335 (147) |

7. Primary Outcome: Elimination Half-life (T1/2) of APR003
Description: as for outcome 2
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 (Cycle duration is 21 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Cohort -1 | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 4 | 0
hr
  Cycle 1 Day 1 | 4.03 (0.816) | 4.56 (1.29) |
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 2 | 0
  Cycle 1 Day 15 | 1.78 (0.630) | 1.77 (0.279) |
  Cycle 2 Day 1: number analyzed (Participants) | 5 | 0 | 0
  Cycle 2 Day 1 | 1.56 (0.485) |  |

8. Primary Outcome: Apparent Volume of Distribution at Steady State After Administration (Vss/F) of APR003
Description: as for outcome 2
Time Frame: Cycle 1 Day 1 (Cycle duration is 21 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Cohort -1 | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 4 | 0
L | 265 (102) | 711 (314) |

9. Primary Outcome: Apparent Total Plasma Clearance (CL/F) of APR003
Description: as for outcome 2
Time Frame: Cycle 1 Day 1 (Cycle duration is 21 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Cohort -1 | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 4 | 0
L/hr | 46.0 (15.7) | 105 (23.1) |

10. Secondary Outcome: Objective Response Rate
Description: Objective response rate (ORR), defined as the proportion of patients with either a complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1
Time Frame: Until disease progression, or up to approximately 15 months and 18 days, whichever is first
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort -1 | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 4 | 1
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Until disease progression, or up to approximately 15 months and 18 days, whichever is first
Groups:
- Cohort -1: 25 MG once weekly
- Cohort 1: 50 MG once weekly
- Cohort 2: 100 MG once weekly
Arm/Group | Cohort -1 | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 3/6 | 1/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/4 | 1/1
Other Adverse Events (participants affected / at risk) | 6/6 | 3/4 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort -1 (N=6) | Cohort 1 (N=4) | Cohort 2 (N=1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) — Dose Limiting Toxicity (DLT)
Progression of Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Post-surgical Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort -1 (N=6) | Cohort 1 (N=4) | Cohort 2 (N=1)
Chills (General disorders) | 5 | 3 | 0
Fever (General disorders) | 2 | 2 | 0
Intermittent fever (General disorders) | 3 | 1 | 0
Fatigue (General disorders) | 3 | 1 | 0
Left chest wall discomfort (General disorders) | 1 | 0 | 0
Intermittent low grade fever (General disorders) | 1 | 0 | 0
Intermittent fatigue (General disorders) | 1 | 0 | 0
Increase thirst (General disorders) | 1 | 0 | 0
Intermittent fever (General disorders) | 0 | 1 | 0
Intermittent generalized body aches (General disorders) | 0 | 1 | 0
Rigors (General disorders) | 1 | 0 | 0
Intermittent chills (General disorders) | 1 | 0 | 0
Edema bilateral lower extremities (General disorders) | 1 | 0 | 0
Intermittent body aches (General disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 2 | 0
Vomiting (Gastrointestinal disorders) | 5 | 1 | 0
Vomiting Intermittent (Gastrointestinal disorders) | 0 | 1 | 0
Nausea Intermittent (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (gas) (Gastrointestinal disorders) | 1 | 0 | 0
Dark colored diarrhea (Gastrointestinal disorders) | 0 | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 3 | 0 | 0
Emesis (Gastrointestinal disorders) | 1 | 0 | 0
Worsening diarrhea (Gastrointestinal disorders) | 0 | 0 | 1
Stomach cramps (Gastrointestinal disorders) | 1 | 0 | 0
Xerostomia (Gastrointestinal disorders) | 0 | 0 | 1
Mouth sores (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Left upper quadrant abdominal discomfort following meals (Gastrointestinal disorders) | 1 | 0 | 0
Intermittent abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Epigastric apin (Gastrointestinal disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Intermitten flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Left flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intermittent right flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intermittent myalgias (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bilateral flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Worsening lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Intermittent anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Anemia of chronic disease (Blood and lymphatic system disorders) | 0 | 1 | 0
Positive COVID-10 test (symptomatic) (Infections and infestations) | 1 | 0 | 0
Bacterial sinusitis (Infections and infestations) | 1 | 0 | 0
Bladder infection (Infections and infestations) | 1 | 0 | 0
Left lower extremity cellulitis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Oral thrush (Infections and infestations) | 0 | 0 | 1
Left upper extremity ringworm (Infections and infestations) | 1 | 0 | 0
Chronic UTI (Infections and infestations) | 0 | 0 | 1
Fever blisters on lower lip (Infections and infestations) | 0 | 1 | 0
Elevation of creatinine (Investigations) | 3 | 0 | 0
Weight loss (Investigations) | 3 | 0 | 0
Intermittent elevation of alkaline phosphatase (Investigations) | 1 | 0 | 0
Elevated alanine transaminase (Investigations) | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0
AST increased (Investigations) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion right lung (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Residual dry cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 1 | 1
Seasonal allergies (Immune system disorders) | 0 | 1 | 0
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Worsening of colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intermittent tumor pain in RUQ/LUQ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intermittent lower abdominal tumor pain flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lower abdominal tumor flare pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Right-sided pleuritic chest tumor flare reaction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Right upper quadrant tumor pain flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumor pain flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rash-face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Diaphoresis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperpigmentation of bilateral fingernails (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 1 | 1 | 0
Worsening hypertension (Vascular disorders) | 1 | 0 | 0
Intermittent hypotension (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 0
Worsening peripheral neuropathy (Nervous system disorders) | 0 | 0 | 1
Persistent change of taste (Nervous system disorders) | 1 | 0 | 0
Lightheadedness (Nervous system disorders) | 1 | 0 | 0
Left hydronephrosis (Renal and urinary disorders) | 2 | 0 | 0
Left ureteral wall thickening (Renal and urinary disorders) | 1 | 0 | 0
Right hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Intermittent dysuria (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0
Intermittent bilateral renal colic (Renal and urinary disorders) | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Worsening diabetes mellitus type 2 (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Post surgical pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hyperbilirubinemia (blood bilirubin increased) (Hepatobiliary disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The primary limitation of this study was its small sample size. While it is difficult to draw firm conclusions on such a small cohort of patients, several preliminary conclusions can be drawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the multicenter publication or 12 months after completion of the Study, whichever occurs first, Institution may itself publish the results of its data from the Study. Institution/Principal Investigator shall provide Sponsor/CRO with advance copy of any proposed publication/oral presentation sixty (60) days prior to the planned date of submission/presentation; Sponsor shall have 60 days to review the proposed publication/presentation.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT04645797/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT04645797/ICF_001.pdf